CLINICAL TRIAL: NCT04910009
Title: The Effect of Privacy Education on Nursing Students' Privacy Consciousness and Attitudes Towards Patient Privacy: A Randomized Controlled Study
Brief Title: The Effect of Privacy Education on Nursing Students' Privacy Consciousness and Attitudes Towards Patient Privacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zehra Göçmen Baykara, Professor, Gazi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2019-252
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Education
Keywords: privacy education; nursing students; privacy consciousness; patient privacy attitudes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Theoretical training group (No Intervention): Students participating in only theoretical training of the privacy education for two 40-minute sessions.
- Digital story and ethical case analysis group (Experimental): Students participating in 2 sessions of 40-minute theoretical training and then participating in 4 sessions of 60-minute digital story and ethical case analysis preparation and presentation.
  Interventions: Other: Four sessions of practical privacy education
- Only ethical case analysis group (Experimental): Students participating in 2 sessions of 40 minutes of theoretical training and then participating in 4 sessions of 60-minute ethical case analysis preparation and presentation only.
  Interventions: Other: Four sessions of practical privacy education

INTERVENTIONS:
Other: Four sessions of practical privacy education — Two sessions of theoretical, four sessions of practical privacy education
  Arms: Digital story and ethical case analysis group; Only ethical case analysis group

SUMMARY:
This study was conducted in a pre-test-post-test, factorial group randomized controlled experimental design to determine the effect of privacy education on nursing students' privacy consciousness and attitudes towards patient privacy. The universe of the study consisted of the third-grade students (n = 239) registered in Gazi University Faculty of Health Sciences Nursing Department in the Fall Semester of the 2020-2021 Academic Year. All students (n = 239) were evaluated according to the exclusion criteria from the study. The students who met the inclusion criteria (n = 116) were informed about the research. A pre-test was applied to the students (n = 116) who volunteered to participate in the study. According to gender, 116 students were randomly assigned to the control group (n = 38), study group I (n = 40), and study group II (n = 38) by a statistician by computer technique. Data were collected November 2020 and February 2021 using the Informative Features Form, the Privacy Consciousness Scale, The Patient Privacy Scale, and Students' Views on Education Form.

DETAILED DESCRIPTION:
Implementation All students participated to the theoretical classes of the privacy education.Theoretical lessons consisted of 2 sessions of 40 minutes each. Privacy Concept and Patient Privacy Specific to Nursing Profession in the first session; In the second session, Ethical Problem Clusters Regarding Patient Privacy in Nursing Practices and Ethical Analysis of Measures to be Taken were explained. In the theoretical sessions, Microsoft PowerPoint presentation, lecture and question-answer methods were used. Then study group I and study group II are divided into four groups. The groups, under the consultancy of the researcher, separately wrote cases involving ethical problems related to physical, informational, decisional, and relational privacy. Both groups made the ethical analysis of these cases into a presentation. The study group I prepared digital storytelling for each case as I extra. The counseling given to the study groups consisted of 2 sessions of 2 hours each. Then, each study groups presented their cases and case studies to their group friends. The study group I shared their digital stories in addition to the case study. Two sessions of 60 minutes each were held for each study group. Two groups made their presentations at each session. Question-answer and discussion methods were used.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Nursing Ethics course for the first time.
* Be a volunteer.

Exclusion Criteria:

* To take the Nursing Ethics Course from a lower class or to be a repeat student,
* Having difficulty in understanding and speaking Turkish (being a foreign national, etc.),
* Graduating from a secondary or higher education institution related to Health Sciences (Nursing, Emergency Medical Technician, Physiotherapy, etc.),
* Not having a computer of his own,
* To report that they have less than intermediate internet access.

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Privacy Consciousness on the 5 mean point The Privacy Consciousness Scale (PCS) Week 8, Week 12, and Week 24 | Baseline, Week 8, Week 12, and Week 24
  The PCS is a validated, self-reported instrument assessing average privacy consciousness. Possible score range from (0) low privacy consciousness to (5) high privacy consciousness
Change from Baseline in Attitudes Toward Patient Privacy on the 5 mean point The Patient Privacy Scale (PPS) Week 8, Week 12, and Week 24 | Baseline, Week 8, Week 12, and Week 24
  The PPS is a validated, self-reported instrument assessing average attitude toward patient privacy. Possible score range from (0) low attitude toward patient privacy to (5) high attitude toward patient privacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Göçmen Baykara, Principal Investigator — Gazi Üniversitesi Sağlık Bilimleri Fakültesi
Locations (1):
- Gülcan Eyüboğlu, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No